CLINICAL TRIAL: NCT06485284
Title: El Camino: Tier 2 Rigorous Evaluation of Promising Interventions in Promotion of Healthy Adolescence
Brief Title: Evaluating the El Camino Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Child Trends (Other)
Collaborators: Identity, Inc. (Unknown); University of Maryland (Other)
Responsible Party: Principal Investigator, Jennifer Manlove, Senior Research Scholar, Child Trends
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TP2AH000077
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Sexual Behavior; Adolescent Behavior
MeSH Terms: conditions — Sexual Behavior; Adolescent Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- El Camino (Experimental): Adolescents receiving the intervention/treatment - El Camino.
  Interventions: Behavioral: El Camino
- Control (Other): Adolescents receiving the control - alternative life skills program.
  Interventions: Behavioral: Life skills program

INTERVENTIONS:
Behavioral: El Camino — El Camino is a goal-setting sexual health promotion program. El Camino's lessons and activities:
  * Are anchored in sexual health promotion and goal-setting
  * Incorporate a goal achievement model throughout the curriculum
  * Are designed with a focus on the needs of Latino youth
  * Focus on the most effective forms of contraception, including long-acting reversible contraceptives
  The El Camino curriculum contains eleven 45-minute lessons and is divided into three sections, or arcs. The three arcs focus on goal setting, sexual and reproductive health, and healthy relationships.
  Arms: El Camino
Behavioral: Life skills program — Youth enrolled in the control condition will receive one of several curricula focused on life skills or leadership, depending on the site and implementation period. These curricula include PODER, an 11-session curriculum that focuses on youth leadership development; Youth Encuentros, a psychoeducational curriculum focused on mental health; El Joven Noble, a youth leadership curriculum; and Courageous Queens, a socio-emotional and character strengthening curriculum.
  Arms: Control

SUMMARY:
The goal of this randomized controlled trial is to evaluate the impacts of El Camino, a goal-setting sexual health promotion program targeted toward Latino adolescents. The primary research questions are:

* Research Question 1: Is participation in the El Camino goal setting program associated with greater abstinence (measured as never had sex, no recent sexual activity) relative to a comparison group that did not receive El Camino?
* Research Question 2: Is participation in El Camino associated with reduced unprotected sex (measured as sex without any method of contraception, sex without a condom) for the intervention group relative to the comparison group?

Researchers will compare those who received El Camino to a comparison group who received an alternative program that does not include sexual health components.

As part of the study, participants will be asked to:

* Attend approximately 11 hours of programming completed over 11 weeks
* Complete baseline, post-intervention, and 12-month follow-up surveys
* For select participants who received the El Camino program, participate in an optional focus group discussion

ELIGIBILITY:
Inclusion Criteria:

* High school student in Montgomery County, MD
* Have not previously received El Camino during pilot study
* Have parental consent (if under 18)
* Agree to be in study

Exclusion Criteria:

* Previously participated in pilot study and received El Camino curriculum
* No parental consent (if under 18)
* Do not agree to be in study

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 746 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Ever had penis-in-vagina sex | Immediately following program completion, 12 months after program completion
  Ever had penis-in-vagina sex (yes/no). Dichotomous variable coded 1 if yes, 0 if no and missing otherwise
Had penis-in-vagina sex in the last three months | Immediately following program completion, 12 months after program completion
  Had penile-vaginal sex in the past three months, even once (yes/no). Dichotomous variable coded 1 if yes, 0 if no and missing otherwise
Had penis-in-vagina sex in the last three months without any method of contraception | Immediately following program completion, 12 months after program completion
  Survey measure: "In the past 3 months, how often have you or your partner used any method of birth control, including condoms, during penis-in-vagina sex?" 5 response categories: 4-point scale from "All of the time" (4) to "None of the time" (1) and I don't know. Coded as 0 if answer is "All of the time". Otherwise coded as 1
Had penis-in-vagina sex in the last three months without use of a condom | Immediately following program completion, 12 months after program completion
  Survey measure: "In the past 3 months, how often have you or your partner used condoms during penis-in-vagina sex?" 5 response categories: 4-point scale from "All of the time" (4) to "None of the time" (1) and I don't know. Coded as 0 if answer is "All of the time". Otherwise coded 1

SECONDARY OUTCOMES:
Intend to use condoms | Immediately following program completion, 12 months after program completion
  Intend to use condoms if having sex (dichotomous variable coded as 1 if responds yes definitely vs. 0 if probably yes, probably not, or
  definitely not)
Intend to use contraception | Immediately following program completion, 12 months after program completion
  Intend to use contraception if having sex (dichotomous variable coded as 1 if responds yes definitely vs. 0 if any other response)
Awareness of birth control methods | Immediately following program completion, 12 months after program completion
  Sum the # of methods responding "yes" to "have you heard of any of these methods of birth control" - response options: 0-6
Knowledge about condoms | Immediately following program completion, 12 months after program completion
  Sum the # of correct responses to 5 items (sample item: "Condoms have an expiration date"-"don't know" is considered an incorrect response)
Knowledge about birth control | Immediately following program completion, 12 months after program completion
  Sum the # of correct responses to 4 items (sample item: "The IUD is more effective at preventing pregnancy than the condom"-"don't know" is considered an incorrect response)
Knowledge about consent | Immediately following program completion, 12 months after program completion
  Sum the # of correct responses to 5 items (sample item: "Is someone consenting to have sex with you if they make out with you clothed"-"don't know" is considered an incorrect response)
Attitudes about birth control | Immediately following program completion, 12 months after program completion
  Average score of 2 items (birth control pills are effective at preventing pregnancy, birth control has too many side effects). Response options on 4-point scale from Strongly disagree to strongly agree)
Attitudes about condoms | Immediately following program completion, 12 months after program completion
  Dichotomous variable measuring 1 if answers "strongly agree" to condoms should always be used, and "strongly disagree" to it is ok if you forget to
  use condoms sometimes. Response options on 4-point scale from Strongly disagree to strongly agree
Definitely know where to get birth control | Immediately following program completion, 12 months after program completion
  Dichotomous variable measured as 1 if respond "definitely" and 0 for all other responses (probably do, probably don't, or definitely don't know where to get birth control methods)
Confidence going to a clinic to get contraception | Immediately following program completion, 12 months after program completion
  Response options on 4-point scale
  from "not at all confident" to
  "completely confident"
Confidence discussing sex, contraception | Immediately following program completion, 12 months after program completion
  Average score of 2 items (how confident you could talk to your partner about whether to have sex, talk to your partner about using condoms. Response options on 4-point scale from "Strongly disagree to strongly agree)
Confidence limit setting | Immediately following program completion, 12 months after program completion
  Average score of 3 items (sample item: "how confident you could say no to sex if your partner won't use a condom") Response options on 4-point scale from "Strongly disagree to strongly agree)
Confidence stating and asking for consent | Immediately following program completion, 12 months after program completion
  Dichotomous variable coded as 1 if "completely confident" on 2 items (vs.
  all other responses)
Decreased psychological distress | Immediately following program completion, 12 months after program completion
  Kessler Psychological Distress Scale (K6) - frequency of 6 symptoms over the past 30 days. Response options on 5-point scale from "none of the time" (coded 1) to "all of the time" (coded 5). Scores summed across all 6 symptoms. Used as a continuous score
Increased educational goal setting | Immediately following program completion, 12 months after program completion
  How likely is it that you will do each of the
  following: (a) graduate from high school; (b) continue education after high school; (c) graduate from college. Response options on a 5-point scale from "not at all likely" (coded 1) to "completely likely" (coded 5). Scores for each item used separately as continuous scores

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Identity, Inc., Gaithersburg, Maryland
  - Montgomery County Public Schools, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faccio B, McClay A, McConnell K, Gates C, Finocharo J, Tallant J, Martinez V, Manlove J. Comparing Virtual and In-Person Implementation of a School-Based Sexual Health Promotion Program in High Schools with Large Latino Populations. Prev Sci. 2023 Dec;24(Suppl 2):251-261. doi: 10.1007/s11121-023-01526-0. Epub 2023 Jun 23. PMID 37351668
- [Derived] McConnell K, Ibrahimi S, Yumiseva M, Shan S, Lewin A. Short-Term Impacts of a School-Based Teen Pregnancy Prevention Program for Latino Youth: a Cluster Randomized Trial. Prev Sci. 2025 Jul;26(5):716-726. doi: 10.1007/s11121-025-01805-y. Epub 2025 Apr 14. PMID 40229508